CLINICAL TRIAL: NCT05251948
Title: A Phase Ib/II, Open-Label, Multicenter, Randomized Umbrella Study Evaluating the Efficacy and Safety of Multiple Treatment Combinations in Patients With Gastric or Gastroesophageal Junction Carcinoma (MORPHEUS C-Gastric and Gastroesophageal Junction Carcinoma)
Brief Title: An Umbrella Study Evaluating the Efficacy and Safety of Multiple Treatment Combinations in Patients With Gastric or Gastroesophageal Junction Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO43408
Record Dates: First submitted 2022-02-09; First posted 2022-02-23 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Gastric and Gastroesophageal Junction Carcinoma
MeSH Terms: interventions — atezolizumab; Capecitabine; Oxaliplatin; Tiragolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atezo + CAPOX (capecitabine + oxaliplatin) (Active Comparator): Participants in the atezolizumab plus capecitabine plus oxaliplatin in Stage 1 will receive treatment until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab; Drug: Capecitabine; Drug: Oxaliplatin
- Atezo + CAPOX +Tira (Experimental): Participants in the atezolizumab plus capecitabine plus oxaliplatin plus tiragolumab arm in Stage 1 will receive treatment until unacceptable toxicity or loss of clinical benefit as determined by the investigator.
  Interventions: Drug: Atezolizumab; Drug: Capecitabine; Drug: Oxaliplatin; Drug: Tiragolumab

INTERVENTIONS:
Drug: Atezolizumab — Atezolizumab is administered by IV infusion on Day 1 of each 21 day cycle. Treatment until progressive disease.
  Other Names: Tecentriq
Drug: Capecitabine — Capecitabine is administered orally twice daily on Days 1-14 of each 21 day cycle. Treatment for up to six cycles.
Drug: Oxaliplatin — Oxaliplatin is administered by IV infusion on Day 1 of each 21 day cycle. Treatment for up to six cycles.
Drug: Tiragolumab — Tiragolumab is administered by IV infusion on Day 1 of each 21 day cycle.
  Arms: Atezo + CAPOX +Tira

SUMMARY:
This is a Phase Ib/II, open-label, multicenter, randomized umbrella study in participants with advanced gastric carcinoma (GC) or gastroesophageal junction carcinoma (GEJC). The study is designed with the flexibility to open new treatment arms as new treatments become available, close existing treatment arms that demonstrate minimal clinical activity or unacceptable toxicity, and modify the participant population. Cohort 1 will enroll participants with inoperable locally advanced, metastatic, or advanced GC or GEJC, with adenocarcinoma confirmed as the predominant histology, who have not received prior systemic therapy for advanced or metastatic disease. Eligible participants will initially be randomly assigned to one of treatment arms (Stage 1). Participants who experience loss of clinical benefit or unacceptable toxicity during Stage 1 may be eligible to receive treatment with a different treatment combination (Stage 2). When a Stage 2 treatment combination is available, this will be introduced by amending the protocol.

ELIGIBILITY:
Inclusion Criteria for Stage 1:

* ECOG Performance Status of 0 or 1
* Inoperable locally advanced, metastatic, or advanced GC or GEJC, with adenocarcinoma confirmed as the predominant histology
* No prior systemic treatment for advanced or metastatic disease
* Life expectancy >= 3 months, as determined by the investigator
* Human epidermal growth factor receptor 2 (HER2)-negative tumors
* Measurable disease according to RECIST v1.1
* Adequate hematologic and end-organ function
* Patients without hepatitis B virus (HBV) infection at screening
* Negative hepatitis C virus (HCV) antibody test at screening, or positive HCV antibody test followed by a negative HCV RNA test at screening
* Negative HIV test at screening
* For women of childbearing potential: agreement to remain abstinent or use contraception, and agreement to refrain from donating eggs, as outlined for each specific treatment arm
* For men: agreement to remain abstinent or use contraception, and agreement to refrain from donating sperm, as outlined for each specific treatment arm

Exclusion Criteria for Stage 1:

* Prior treatment with CD137 agonists or immune checkpoint blockade therapies
* Treatment with investigational therapy within 28 days prior to initiation of study treatment
* Any contraindications to any of the study drugs of the chemotherapy regimen
* Eligible only for the control arm
* Patients with a signet ring cells dominant carcinoma
* Symptomatic, untreated, or actively progressing CNS metastases
* History of leptomeningeal disease
* Active or history of autoimmune disease or immune deficiency
* Significant cardiovascular disease within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
* History of malignancy other than GC or GEJC within 2 years prior to initiation of study treatment, with the exception of malignancies with a negligible risk of metastasis or death

Exclusion Criteria for Tiragolumab-Containing Arm:

* Prior treatment with an anti-TIGIT agent
* Active Epstein-Barr virus (EBV) infection or known or suspected chronic active EBV infection at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-09-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 3-5 years
  ORR is defined as the proportion of participants with a complete response or a partial response on two consecutive occasions >= 4 weeks apart during Stage 1, as determined by the investigator according to RECIST v1.1.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Randomization to the first occurrence of disease progression or death from any cause (whichever occurs first) (up to approximately 3-5 years)
  PFS after randomization is defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first) in Stage 1, as determined by the investigator according to RECIST v1.1.
Overall Survival (OS) | Randomization to death from any cause (up to approximately 3-5 years)
  OS after randomization, defined as the time from randomization to death from any cause, regardless of stage.
Overall Survival (OS) | At specific timepoints (up to approximately 3-5 years)
  OS at specific timepoints.
Duration of Response (DOR) | First occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first) (up to approximately 3-5 years)
  DOR is defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first) in Stage 1, as determined by the investigator according to RECIST v1.1.
Disease Control Rate | Up to approximately 3-5 years
  Disease control rate is defined as the proportion of participants with stable disease for >= 12 weeks or a complete or a partial response, as determined by the investigator according to RECIST v1.1.
Percentage of Participants with Adverse Events in Stage 1 | Baseline through approximately end of study (approximately 3-5 years)
  Percentage of participants with adverse events in Stage 1.
Percentage of Participants with Adverse Events in Stage 2 | Baseline through approximately end of study (approximately 3-5 years)
  Percentage of participants with adverse events in Stage 2.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- China (12):
  - The General Hospital of People?s Liberation Army (301 Hospital), Beijing
  - the First Hospital of Jilin University, Changchun
  - First Affiliated Hospital of Gannan Medical University, Ganzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Sir Run Run Shaw Hospital, School of Medicine, Zhejiang University, Hangzhou
  - The Second Affiliated Hospital of Anhui Medical University, Hefei
  - Affiliated Hopsital of Jining Medical University, Jining
  - Nanjing Drum Tower Hospital, the Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Nan Tong Tumor Hospital, Nantong
  - Shanxi Province Cancer Hospital, Taiyuan
  - The First Affiliated Hospital of Xian Jiao Tong University, Xi'an
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing